CLINICAL TRIAL: NCT03183284
Title: Comparison Study of Methyl Prdnisolone Versus Intravenous Dexamethazone in Severe Immune Thrombocytopenic Purpra
Brief Title: Comparison Between Methyl Prednisolone and Intravenous Dexamethazone in Severe Immune Thrombocytopenic Purpra
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hager mohammed, assiut, Assiut University
Other Study IDs: Hager2791
Record Dates: First submitted 2017-05-14; First posted 2017-06-12 (Actual); Last update posted 2017-06-12 (Actual); Status verified 2017-06

CONDITIONS: Immune Thrombocytopenia
Keywords: dexamethazone; prednislone; severe ITP
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Immune thrombocytopenic purpra(ITP) is an autoimmune thrombocytopenic syndrome characterized by decreased platelet count and increased risk of bleeding, primarily due to immunoglobulins G(IgG)autoantibodies opsonizing the individual's platelets,resulting in markedly enhanced Fc receptors(FcR)-mediated phagocytosis and destruction by macrophages in the reticuloendothelial system within spleen Severe ITP defined as :Patients who have clinically relevant bleeding that mean that patients have bleeding symptoms at presentation sufficient to mandate treatment,or occurrence of new bleeding symptoms requiring additional therapeutic intervention with a different platelet-enhancing agent or an increased dose.

DETAILED DESCRIPTION:
Immune thrombocytopenic purpra(ITP) is an autoimmune thrombocytopenic syndrome characterized by decreased platelet count and increased risk of bleeding, primarily due to immunoglobulins G(IgG)autoantibodies opsonizing the individual's platelets,resulting in markedly enhanced Fc receptors(FcR)-mediated phagocytosis and destruction by macrophages in the reticuloendothelial system within spleen Severe ITP defined as :Patients who have clinically relevant bleeding that mean that patients have bleeding symptoms at presentation sufficient to mandate treatment,or occurrence of new bleeding symptoms requiring additional therapeutic intervention with a different platelet-enhancing agent or an increased dose.Prednislone is the standard intial first-line therapy in naïve ITP patients.Prednislone is usually given at 0.5 to 2mg/kg until platelet count increase(>30-50 *10^9/L )which may require several days to several weeks,however prednisone should be rapidly tapered after 4 weeks to avoid corticosteroid related complication. In a trial to shorten the duration and reduce adverse effects of corticosteroids treatment. Dexamethasone in a dose of 40mg/day has been administered for 4days (equivalent to~400mg of prednisone per day) achieved 85% initial reponse and sustained response 50% of adult cases of ITP at 6 months follow up

ELIGIBILITY:
Inclusion Criteria:

* Patients were aged 18or older diagnosed as acute severe ITP presented with active bleeding for emergency treatment.

Exclusion Criteria:

* Any contraindications for steroid therapy (osteoprosis, uncontrolled diabetes or uncontrolled hypertension).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients will be recruited in each group of therapy IV dexamethasone 40 mg/ day for 4 days versus IV methyl prednisolone 1 gm/day for 3 days.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-06-30 (Estimated); Primary Completion 2017-06-30 (Estimated); Study Completion 2018-06-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients respond to intravenous dexamethazone compared to patients received intravenous methylprednisolone in severe immune thrombocytopenic purpra | one year

IPD SHARING:
Plan to Share IPD: No